CLINICAL TRIAL: NCT01659476
Title: Bronchodilating and Bronchoprotective Effects of Deep Inspirations in Asthma, Cough Variant Asthma and Chronic Cough With Normal Airway Sensitivity and Sensory-Mechanical Responses to High-Dose Methacholine in Healthy Normal Subjects
Brief Title: Bronchodilating and Bronchoprotective Effects of Deep Inspirations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Diane Lougheed, MD, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2012-01
Record Dates: First submitted 2012-07-30; First posted 2012-08-07 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Asthma; Cough
Keywords: methacholine; deep inspiration; bronchoprotective effect; bronchodilating effect
MeSH Terms: conditions — Asthma; Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Asthma (Experimental): Individuals diagnosed with asthma.
  Interventions: Other: Methacholine(MCh) Challenge Testing
- Cough Variant Asthma (Experimental): Individuals diagnosed with cough variant asthma.
  Interventions: Other: Methacholine(MCh) Challenge Testing
- Mch-induced cough w/normal airway sensitivity (Experimental): Individuals with chronic cough normal PC20 MCh(>16 mg/mL) & who cough during Mch challenge testing.
  Interventions: Other: Methacholine(MCh) Challenge Testing
- Normal (Experimental): Individuals with no history of asthma or chronic cough
  Interventions: Other: Methacholine(MCh) Challenge Testing

INTERVENTIONS:
Other: Methacholine(MCh) Challenge Testing — Visit 1: High-dose methacholine challenge test
  Visit 2 or 3: Will be conducted in random order and subjects will perform one of two modified single-dose methacholine challenge tests at either visit. During these modified challenges, subjects will (a) perform five DIs from functional residual capacity (FRC) to total lung capacity (TLC) back to FRC, or (b) refrain from taking DIs prior to inhaling the previously measured single PC20 dose of methacholine.
  Other Names: Drug:MCh[inhalation of sequential doubling doses of MCh(0.0625-256 mg/mL)]; Other names: Provocholine
  Arms: Asthma; Cough Variant Asthma; Mch-induced cough w/normal airway sensitivity
Other: Methacholine(MCh) Challenge Testing — Visit 1: Baseline tests, and subjects will be randomized to complete either a high-dose methacholine using maximal expiratory flow-volume loop (MEFV), or a high-dose methacholine challenge with impulse oscillometry (IOS) and partial expiratory flow-volume loop (PEFV) and MEFV at each dose step.
  Visit 2: Subjects will perform the opposite protocol, based on their first visit:
  Other Names: Drug:MCh[inhalation of sequential doubling doses of MCh(0.0625-256 mg/mL)]; Other names: Provocholine
  Arms: Normal

SUMMARY:
The objectives of this research are to compare (i) the bronchodilating and (ii) the bronchoprotective effects of deep inspirations (DIs) in individuals with: (a) asthma, (b) CVA, (c) methacholine-induced cough but normal airway sensitivity and .

(d) in healthy individuals (without asthma, chronic cough or asymptomatic airway hyperresponsiveness).

Hypotheses:

i. The bronchodilating effect of a DI will be: (a) absent or impaired in individuals with classic asthma; (b) impaired in individuals with CVA; (c) preserved in individuals with methacholine-induced cough but normal airway sensitivity; and (d) preserved in healthy individuals (without asthma, chronic cough or asymptomatic airway hyperresponsiveness).

ii. The bronchoprotective effect of a DI will be: (a) absent in individuals with classic asthma; (b) impaired in individuals with CVA; (c) preserved in those with methacholine-induced cough but normal airway sensitivity; and (d) preserved in healthy individuals (without asthma, chronic cough or asymptomatic airway hyperresponsiveness).

iii. Healthy individuals without asthma, chronic cough, or asymptomatic airway hyperresponsiveness, will not cough, or develop significant dyspnea, small airways obstruction or dynamic hyperinflation during high-dose methacholine bronchoprovocation.

DETAILED DESCRIPTION:
Asthma is a chronic respiratory condition characterized by eosinophilic airway inflammation. Individuals with classic asthma experience paroxysmal symptoms including cough, wheeze, shortness of breath and chest tightness. Cough variant asthma (CVA) is asthma in which chronic cough (cough lasting eight weeks or more) is the sole or predominant symptom of asthma. The pathophysiologic mechanisms which differentiate asthma, CVA, and eosinophilic bronchitis without asthma are not fully understood. We have recently identified individuals with chronic cough who cough during methacholine but have normal airway sensitivity (ie. do not have asthma or CVA) and may or may not have eosinophilic bronchitis. The purpose of this research is to examine the pathophysiologic differences between three causes of chronic cough: asthma, cough variant asthma and methacholine-induced cough with normal airway sensitivity. The responses in healthy normal subjects are crucial to understand the clinical relevance of methacholine-induced cough with normal airway sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-65 years of age with asthma, CVA and individuals with methacholine-induced cough but normal airway sensitivity. The following definitions will be used:

  1. asthma: episodic respiratory symptoms occurring in association with variable airflow obstruction (Canadian Asthma Consensus Report definition);
  2. CVA: chronic cough (≥8 weeks) is the sole or predominant symptom and positive methacholine challenge (PC20 ≤ 16 mg/mL) and history of cough responding to specific asthma treatment (such as inhaled steroid or 1 week trial of bronchodilator);
  3. Methacholine-induced cough but normal airway sensitivity: chronic cough (≥8 weeks) is the sole or predominant symptom and negative methacholine challenges (PC20 > 16 mg/mL).
* Individuals aged 18-65 years of age with no history of asthma or chronic cough.

Exclusion Criteria:

* an exacerbation necessitating a change in medication, emergency department visit or hospitalizations within the previous 4 weeks
* inability to perform acceptable spirometry
* medical contraindications to methacholine challenge testing

  1. Severe airflow limitation (FEV1 <50% predicted or <1.0 L);
  2. Heart attack or stroke in last 3 months;
  3. Uncontrolled hypertension, systolic BP > 200 or diastolic BP > 100;
  4. Known aortic aneurysm;
  5. Moderate airflow limitation <60% predicted or 1.5) is a relative contraindication;
  6. Inability to perform acceptable quality spirometry;
  7. Current use of cholinesterase inhibitor medication (for myasthenia gravis); and
  8. Pregnant or nursing mothers.
* smoking history in excess of 10 pack years

Note: Previous treatment with inhaled or systemic corticosteroids is not an exclusion criterion; medication use will be recorded and examined in the analysis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-10; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Mid expiratory flows | Time frame of the methacholine challenge varies between individuals. At provocative concentration of methacholine causing a 20% and 50% decline in FEV1 (PC20 and PC50 respectively). On average, these occur about 15-25 minutes into the challenge test.
  The bronchodilating effect of a DI will be examined using responses to high-dose methacholine challenge testing (Visit 1) in these subgroups by comparing the mid-expiratory flow difference between the partial (PEF) and full maximal flow-volume (MEF) loops at 40% above Residual Volume (RV) from the forced vital capacity (FVC) (PEF40 and MEF40 respectively) at PC20 and PC50 with that recorded at baseline.

SECONDARY OUTCOMES:
percent fall in FEV1 | After methacholine administration; will occur 2-5 minutes after 1 dose of methacholine.
  The bronchoprotective effect of a deep inspiration will be measured by the difference between the percent fall in FEV1 following administration of methacholine using modified single-dose methacholine challenge tests on Visits 2 and 3 (with or without preceding deep inspirations)
respiratory system reactance (X5) | After methacholine administration; will occur 2-5 minutes after 1 dose of methacholine.
  The bronchoprotective effect of a DI will be also examined by comparing mechanical responses to methacholine using impulse oscillometry (IOS). Single IOS will measure peripheral airway function using respiratory system reactance (X5) and peripheral resistance (R5-R20) and central resistance (R20) will be used as an index of airway narrowing.
peripheral resistance (R5-R20) | After methacholine administration; will occur 2-5 minutes after 1 dose of methacholine.
  The bronchoprotective effect of a DI will be also examined by comparing mechanical responses to methacholine using impulse oscillometry (IOS). Single IOS will measure peripheral airway function using respiratory system reactance (X5) and peripheral resistance (R5-R20) and central resistance (R20) will be used as an index of airway narrowing.
Central airway resistance | After methacholine administration; will occur 2-5 minutes after 1 dose of methacholine.
  The bronchoprotective effect of a DI will be also examined by comparing mechanical responses to methacholine using impulse oscillometry (IOS). Single IOS will measure peripheral airway function using respiratory system reactance (X5) and peripheral resistance (R5-R20) and central resistance (R20) will be used as an index of airway narrowing.
Forced vital capacity (FVC) | After methacholine administration; will occur 2-5 minutes after 1 dose of methacholine.
  As an index of airway closure.
FEV1/FVC | After methacholine administration; will occur 2-5 minutes after 1 dose of methacholine.
  As an index of airway narrowing (obstruction)

CONTACTS AND LOCATIONS:
Overall Officials: M. Diane Lougheed, MD MSc, Principal Investigator — Queen's University
Locations (1):
- Kingston General Hospital at Queen's University, Kingston, Ontario, Canada